CLINICAL TRIAL: NCT02292849
Title: Peer to Peer Delivery of Behavioral Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1307014080; P30MH085943 (NIH)
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer to Peer (Experimental): These individuals will receive a standard mental health referral to a community agency and in addition meet with a trained peer coach for 12 weekly meetings.
  Interventions: Behavioral: Peer to Peer
- Referral (Active Comparator): These individuals will receive a standard mental health referral to a community agency.
  Interventions: Other: Standard Mental Health Referral

INTERVENTIONS:
Behavioral: Peer to Peer — 12 weekly sessions of peer-delivered behavioral activation
  Arms: Peer to Peer
Other: Standard Mental Health Referral — Standard mental health referral to a community agency
  Arms: Referral

SUMMARY:
The goal of this study is to test the feasibility, acceptability and preliminary impact of peer-delivered Behavioral Activation (BA) for depressed older adults (60+) who are Naturally Occurring Retirement Communities (NORC) residents or senior center participants.

DETAILED DESCRIPTION:
This project focuses on helping to solve a growing problem in health care today. Through increased screening in the older adult population, detection of depression has increased which has established a growing need for mental health resources. Unfortunately, there are limited resources to keep up with the steady increase of individuals in need. Training peers to work with older depressed adults in techniques such as behavioral activation provides an alternative model to help moderate the increased need and provide a unique intervention of care. Developing an innovative peer facilitated program has the potential to enhance the delivery of quality health care.

The specific aims of the study are 1) to train peer coaches and implement Peer to Peer in the community 2) to examine depression ratings over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Member of Lenox Hill Senior Center, St. Peter's Senior Center, or Beth Abe
* Score of 10+ on Patient Health Questionnaire (PHQ-9)

Exclusion Criteria:

* Presence of alcohol abuse, substance abuse, psychotic disorder, or bipolar disorder as observed on the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID)
* Inability to speak English
* Dementia: Mini Mental State Examination (MMSE) score below 24
* High suicide risk, i.e. intent or plan to attempt suicide

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Raue, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raue PJ, Sirey JA, Dawson A, Berman J, Bruce ML. Lay-delivered behavioral activation for depressed senior center clients: Pilot RCT. Int J Geriatr Psychiatry. 2019 Nov;34(11):1715-1723. doi: 10.1002/gps.5186. Epub 2019 Aug 8. PMID 31368583

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer to Peer Coaches: Peer coaches who were eligible to provide the Behavioral Activation intervention
- Peer to Peer Clients: These individuals will receive a standard mental health referral to a community agency and in addition meet with a trained peer coach for 12 weekly meetings.
  Peer to Peer: 12 weekly sessions of peer-delivered behavioral activation
- Referral Clients: These individuals will receive a standard mental health referral to a community agency.
  Standard Mental Health Referral: Standard mental health referral to a community agency
Period: Overall Study
Arm/Group | Peer to Peer Coaches | Peer to Peer Clients | Referral Clients
Started | 11 | 8 | 10
Completed | 7 | 6 | 8
Not Completed | 4 | 2 | 2
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Physician Decision | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peer to Peer Coaches: These individuals were eligible to provide the Behavioral Activation intervention.
- Total: Total of all reporting groups
Arm/Group | Peer to Peer Coaches | Peer to Peer Clients | Referral Clients | Total
Number analyzed (Participants) | 11 | 8 | 10 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 11 | 8 | 10 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 10 | 24
  Male | 2 | 3 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 11 | 8 | 8 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 7 | 7 | 9 | 23
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Peer to Peer Coaches Who Undergo Behavioral Activation Training and Achieve Certification
Description: Proportion of Peer to Peer coaches who undergo Behavioral Activation training and achieve certification
Time Frame: 4 weeks prior to Baseline
Population: This outcome analyzed Peer to Peer coaches who were eligible to provide the Behavioral Activation intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Peer to Peer Coaches
Number analyzed (Participants) | 11
Participants | 7

2. Primary Outcome: Number of Peer to Peer Clients Who Attend > 80% of Behavioral Activation Sessions
Description: Number of Peer to Peer clients who attend > 80% of Behavioral Activation sessions
Time Frame: 12 weeks
Population: Clients assigned to receive Peer BA
Measure: Count of Participants; unit: Participants
Groups:
- Peer to Peer Clients: Those individuals will receive a standard mental health referral to a community agency and in addition meet with a Peer Coach for 12 weekly meetings.
Arm/Group | Peer to Peer Clients
Number analyzed (Participants) | 8
Participants | 8

3. Secondary Outcome: Changes in Hamilton Depression Rating Scale Scores
Description: Hamilton Depression Rating Scale mean change scores from baseline to 12 weeks. This scale measures severity of depressive symptoms (range=0-76), with higher scores indicating more sever depressive symptomatology.
Time Frame: Baseline and 12 weeks
Population: Randomized clients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer to Peer Clients | Referral Clients
Number analyzed (Participants) | 6 | 8
units on a scale | -8.0 (4.3) | 0.0 (7.5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Peer to Peer Clients | Referral Clients
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer to Peer Clients (N=8) | Referral Clients (N=10)
ER visit for respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ER visit for injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ER visit for general disorder (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No